CLINICAL TRIAL: NCT02885974
Title: Pilot Study of Celecoxib Combined With Gemcitabine and Cisplatin for Neoadjuvant Treatment of Localized, Muscle-Invasive Bladder Cancer
Brief Title: Celecoxib With Chemotherapy in Localized, Muscle-Invasive Bladder Cancer
Acronym: BLAST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Aihua Edward Yen, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-36486
Record Dates: First submitted 2016-05-23; First posted 2016-09-01 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Bladder Cancer
Keywords: Celecoxib; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Celecoxib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (1):
- Celecoxib plus Gemcitabine/Cisplatin chemo (Experimental): Celecoxib plus Gemcitabine/Cisplatin neoadjuvant chemotherapy
  Interventions: Drug: Celecoxib; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Celecoxib — Celecoxib (100 mg daily)
Drug: Gemcitabine — 1,000 mg/m2 (IV), on Days 1 and 8 of each 21-day cycle. Up to 4 cycles.
Drug: Cisplatin — 70 mg/m2 (IV), on Day 1 of each 21-day cycle. Up to 4 cycles.

SUMMARY:
The purpose of this study is to compare patient tumor tissue before and after treatment with chemotherapy plus celecoxib. Investigators will look at gene expression, to see what effect celecoxib may have on tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or their legally authorized representative must be informed of the investigational nature of this study, and must sign and give written informed consent in accordance with institutional and federal guidelines.
* Patients must have histologically proven urothelial carcinoma of the bladder. Those with mixed histology, including a component of urothelial carcinoma, are eligible. Pure small cell carcinoma, pure adenocarcinoma, and pure squamous cell carcinoma are excluded.
* Patients must have Stage cT2-T4a N0 M0 disease. Clinical T stage is based on the TURBT sample, exam under anesthesia and cross-sectional imaging studies. Patients must undergo cystoscopy and TURBT as part of the staging procedure within 120 days prior to registration.

To exclude non-bulky/low-risk tumors, subjects must have documented muscle invasion with at least one of the following:

i. Disease measuring at least 10 mm on cross-sectional imaging. Bladder thickening on imaging, by itself, is not adequate.

ii. The presence of tumor-associated hydronephrosis.

* Patients must have staging scans with abdominal/pelvic CT or MRI scan, and CT scan or x-ray of the chest within 56 days prior to registration. If the alkaline phosphatase is > 1.5 x upper limit of normal (ULN), there is a presence of suspicious bone pain, or if there is other clinical suspicion of bone metastases, a whole body bone scan is required within 56 days prior to registration.
* Patients must have a Zubrod performance status of 0, 1 or 2.
* Patients must be 18 years of age or older.
* Patients must have adequate renal function as evidenced by calculated creatinine clearance ≥ 50 mL/min. The serum creatinine value used in the calculation must have been obtained within 28 days prior to registration.
* Patients must have adequate hepatic function (within 28 days prior to registration), defined as:

  i. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (or ≤ 2.5 x ULN with Gilbert's disease); and ii. SGOT (AST) ≤ 2 x institutional ULN; and iii. SGPT (ALT) ≤ 2 x institutional ULN.
* Patients must have adequate hematologic function (within 28 days prior to registration), defined as:

  i. Absolute neutrophil count (ANC) ≥ 1,500/μL; and ii. Hemoglobin ≥ 9 g/dL; and iii. Platelets ≥ 100,000/μL.
* Patients must have tumor tissues from transurethral resection of the bladder tumor (TURBT) that is within 120 days of registration and available for submission. Tissue sample must be sufficient for IHC testing; that is,it must be sufficient tumor tissues for correlative science after pathologic diagnosis [i.e., enough tumor tissue to pass the staging criteria in 4c].
* Patients must consent to the submission of FFPE blocks and/or unstained slides.

Exclusion Criteria:

* Patients must not have received previous systemic cytotoxic chemotherapy for urothelial carcinoma.
* Patients must not have peripheral neuropathy ≥ Grade 2.
* Patients must not have presence of Class III or IV heart failure, according to New York Heart Association Classifications, or a known left ventricular ejection fraction of less than 50%. Note: LVEF evaluation by echocardiogram or multi-gated acquisition scan (MUGA) is not required prior to registration.
* Patients must not have a significant history of bleeding events. Patients with a history of a significant bleeding episode (e.g. hemoptysis, upper or lower GI bleeding, grade 3 or 4 gross hematuria unable to be controlled by trans-urethral resection of the bladder tumor) within 6 months of registration are not eligible.
* No arterial thrombotic events within 6 months of registration, including transient ischemic attack (TIA), cerebrovascular accident (CVA), peripheral arterial thrombus, unstable angina or angina requiring surgical or medical intervention in the past 6 months, or myocardial infarction (MI). Patients with clinically significant peripheral artery disease (i.e., claudication on less than one block) are ineligible.

Patients who have experienced a deep venous thrombosis or pulmonary embolus within the past 6 months must be on stable therapeutic anticoagulation to be enrolled to this study.

* In the opinion of the treating investigator, the patient must be a candidate to receive gemcitabine/cisplatin treatment.
* Patients must not have aspirin sensitive asthma.
* Patients must not be known to have hypersensitivity to cisplatin, gemcitabine, or celecoxib.
* Patients must not have any incidence of or uncontrolled medical illness (e.g. active cardiac symptoms, active systemic infection, etc.) that would limit the patient's ability to participate in the protocol.
* Patients must not be pregnant or nursing due to the potential teratogenic side effects of the protocol treatment. Women/men of reproductive potential must agree to use an effective contraceptive method during and for 6 months after completing protocol treatment. A negative pregnancy test is required within 7 days prior to registration for women of child-bearing potential.
* Patients are ineligible if they plan on regular use of NSAIDs at any dose more than 2 times per week (on average) or aspirin at more than 325 mg at least three times per week, on average. Low-dose aspirin not exceeding 100 mg/day is permitted. Patients who agree to stop regular NSAIDs or higher dose aspirin are eligible and no wash out period is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-12; Primary Completion 2024-03 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
mRNA expression in pre- and post-chemotherapy tissues | Up to four 21-day cycles of chemotherapy.
Number and severity of adverse events | Until 30 days after last treatment.

SECONDARY OUTCOMES:
Pathological disease stage at cystectomy, including the rate of pT0 and the rate of < pT2. | At surgery, within 70 days after completing chemotherapy
Two-year progression free survival | Up to 2 years
Two-year overall survival | Up to 2 years

OTHER OUTCOMES:
Changes Cytokeratin 14 and phospho-histone H3 (proliferation markers) | Between baseline and treatment completion, up to 154 days
  Correlative Objective
Changes in COX2 IHC staining | Through treatment completion, up to 154 days
  Correlative Objective
Changes in gene expression signatures in association with therapeutic response | Through treatment completion, up to 154 days
  correlative objective

CONTACTS AND LOCATIONS:
Overall Officials: Aihua Edward Yen, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor Clinic, Houston, Texas
  - Harris Health System - Smith Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No